CLINICAL TRIAL: NCT01106560
Title: A Single Centre Prospective Randomised Controlled Clinical Trial Comparing Total Hip Arthroplasty Performed Either Through a Posterior Approach or a Direct Anterior Approach
Brief Title: A Randomised Trial Comparing Anterior Versus Posterior Approach in Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01.004.12 rev.01
Record Dates: First submitted 2010-04-15; First posted 2010-04-20 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

ARMS (2):
- Anterior Approach Group (Active Comparator): (AMIS)
  Interventions: Procedure: Minimally Invasive Anterior Approach
- Posterior Approach Group (Active Comparator): (Posterior)
  Interventions: Procedure: Standard postero-lateral approach

INTERVENTIONS:
Procedure: Minimally Invasive Anterior Approach — Anterior minimally invasive surgery (AMIS)
  Arms: Anterior Approach Group
Procedure: Standard postero-lateral approach
  Arms: Posterior Approach Group

SUMMARY:
This is a single-centre, randomised, prospective clinical follow-up study to evaluate clinical outcome and gait analysis after total hip arthroplasty using the standard postero-lateral approach or the minimally invasive anterior approach.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-75 years at time of surgery.
* Those presenting with primary or secondary osteoarthritis and/or rheumatoid arthritis of the hip.
* Those deemed capable of giving informed consent, understanding the aims of the study and expressing willingness to comply with the post-operative review programme.
* Patients who signed the study consent form prior to surgery.

Exclusion Criteria:

* Pregnant women or women who plan to conceive in the future.
* Those whose prospects for a recovery to independent mobility would be compromised by known coexistent, medical problems.
* Those already treated by with a Total Hip Replacement (THR) (i.e. requiring a revision hip replacement).
* Those with co-existent ipsilateral knee disease or back problems
* Muscle contracture around the hip joint
* Individuals who have undergone organ transplant.
* Those with a known co-existent medical condition where death is anticipated within five years due to the pre-existing medical condition.
* Individuals who have had a THR on the contra-lateral side within the 6 months.
* Individuals who have undergone a THR on the contralateral side and whose outcome is considered unsatisfactory or not good. An unsatisfactory or poor result is defined as achieving a total UCLA score (including activity) < 16 points.
* Individuals requiring bilateral hip replacement.
* Individuals whose body mass index (BMI; kg/m2) >35.
* Individuals with active or suspected infection or sepsis.
* Individuals with renal failure and/or renal insufficiency.
* Patients with severe forms of developmental dysplasia of the hip (DDH): Crowe types II, III, IV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Compare gait kinematics and the return to normalization of gait in patients that have undergone a THA via the direct anterior approach vs. the posterior approach | on average up to 6 weeks

SECONDARY OUTCOMES:
Clinical assessment of patient using the Harris Hip Score | pre-op and 6 weeks, 6 months, 1 year after surgery
Assessment of the improvement in quality of life and joint movement using the EuroQol-5D Score | pre-op, 1 year post-op
Assessment of patient's level of activity using the UCLA score | pre-op and 6 weeks, 6 months, 1 year after surgery
Radiological evaluation to assess the fixation and stability of femoral and acetabular components | pre-op and 6 weeks, 6 months, 1 year after surgery
Strength Testing | 6 weeks, 6 months and 1y after surgery
  Muscle strength will be assessed using the MIE digital myometer (from patient #50 to patient #100)
MRI evaluation | preop-1y after surgery
  A MRI examination will be used to detect any damage in the hip musculature and tendons (from patient #50 to patient #100)
Assessment of gait kinematics | 6 weeks, 12 weeks and 6 months
  Comparison gait analysis Anterior vs Posterior groups at fixed time point (from patient #50 to patient # 100)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Field, PhD FRCS(Orth), Principal Investigator — British Orthopaedic Association
Locations (1):
- The Elective Orthopaedic Centre (EOC), Epsom, United Kingdom